CLINICAL TRIAL: NCT04444375
Title: Plantar Pain, Balance and Foot Function in Individuals With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Duray, Principal Investigator, Suleyman Demirel University
Other Study IDs: 60116787-020/71494
Record Dates: First submitted 2020-05-29; First posted 2020-06-23 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; plantar pain; body mass index; obesity; balance; foot pain; disability
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Recruitment Detection, Audiologic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obese, non-obese: obese and non-obese diabetic patients
  Interventions: Diagnostic Test: balance test

INTERVENTIONS:
Diagnostic Test: balance test — balance test

SUMMARY:
Diabetes Mellitus (DM) and increase of body mass index (BMI) are two one of the most common risk factors for plantar pain and related disability. The aim of our study was to evaluate the relationship between plantar pain, balance and foot function in diabetic DM patients has with different BMI.

ELIGIBILITY:
Inclusion Criteria:

* having plantar pain
* and no change in BMI by more than 10% for at least 3 months
* being volunteer to participate to the study

Exclusion Criteria:

* having musculoskeletal surgery for foot
* having neurological, orthopedic, and cardiovascular diseases
* vision and hearing problems that may cause balance disorder

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Diabetes Mellitus
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
the Portable Computerized Kinesthetic Equilibrium Device (SportKAT 550) | 6 months
  balance
Foot Function Index | 6 months
  Foot Function Index of 23 items, and evaluates the pain, disability and activity limitation. The each of the pain and insufficiency subscales consist of 9 items and the activity limitation subscale includes 5 items. Patients score their foot pain level with Visual Analogue Scale (VAS) in various situations during the last 1 week. To calculate the scores of the index, the score of each item are summed, then divided by possible the maximum score can be obtained from the FFI. Higher scores indicate greater pain, disability and activity limitation level.
Manchester Foot Pain and Disability Index | 6 months
  Manchester Foot Pain and Disability Index consists of 4 subsections including 9 questions for inadequacy, 5 questions for pain, 3 questions for concern and 2 questions for difficulty. Each item is scored between 0-2. The total score is calculated by summing the scores from all items. Higher scores indicate worse health situation.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Duray, Principal Investigator — Suleyman Demirel University
Locations (1):
- Mehmet Duray, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No